CLINICAL TRIAL: NCT00817609
Title: Effectiveness and Safety of Angongniuhuang Pill on Restoring Consciousness for Patients Who Have Suffered From a Stroke
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Office for Traditional Chinese medicine, Shanghai Municipal Health Bureau
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008L060A
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2009-09

CONDITIONS: Stroke; Acute Ischemic Stroke
Keywords: Angongniuhuang Pill; consciousness level of patients who suffered from a stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental)
  Interventions: Drug: Angongniuhuang Pill
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Angongniuhuang Pill — 7 days of Angongniuhuang Pill
  Arms: A
Drug: placebo — 7 days of placebo
  Arms: B

SUMMARY:
This study will determine if Angongniuhuang Pill (Composed of Niuhuang, Yujin, Xijiao, Huangqin, Huanglian, Xionghuang, Zhizi, Zhusha, Bingpian, Shexiang, and Zhenzhu) will have a better effect in restoring consciousness for patients who have suffered from an acute ischemic stroke. The study is designed to look at both consciousness level and overall recovery and recovery of motor function, for example muscle strength and coordination.

ELIGIBILITY:
Inclusion Criteria:

* Occurrence of an acute ischemic stroke (between 9 and 72 h after onset) with
* A score of not higher than 12 of Glasgow Coma Scale (GCS)
* Patient age of between 18 and 80 years.
* Patients or their representatives voluntarily take part in this study and signed the informed consent

Exclusion Criteria:

* Transient Ischemic attack(TIA), cerebral hemorrhage, subarachnoid hemorrhage
* Ischemic stroke that needs rt-PA treatment
* Subjects who are unlikely to complete taking the investigational product and/or are unlikely to undergo active medical management during that period due to a severe clinical condition.
* Pregnant or breast-feeding.
* Proven disability by law, such as blindness, deafness, dumb, disturbance of intelligence, mental disorders, limb handicap.
* Liable to be allergic (allergic to at lease 2 foods/drugs previously exposed)
* Had been participated in other clinical trials during the last 1 month prior to study inclusion.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)

PRIMARY OUTCOMES:
Glasgow Coma Scale (GCS) within 90 days after stroke onset. | 90 days

SECONDARY OUTCOMES:
The percentage of patients of different consciousness level stratified according to the GCS, and the time spent of patients who recovered from coma. | 90 days
Global disability on modified Rankin scale at 90 days. | 90 days
NIH stroke scale | 90 days
Changes in laboratory indexes as safety assessment, including red blood cell(RBC), white blood cell(WBC), platelet(PLT), alanine transarninase(ALT), aspartate transarninase (AST), blood urea nitrogen (BUN), creatinine(Cr) in blood samples; protein, red b | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Tsao JW, Hemphill JC 3rd, Johnston SC, Smith WS, Bonovich DC. Initial Glasgow Coma Scale score predicts outcome following thrombolysis for posterior circulation stroke. Arch Neurol. 2005 Jul;62(7):1126-9. doi: 10.1001/archneur.62.7.1126. PMID 16009770